CLINICAL TRIAL: NCT00059982
Title: Phase II Trial Of Perifosine In Locally Advanced, Unresectable Or Metastatic Pancreatic Adenocarcinoma
Brief Title: Perifosine in Treating Patients With Locally Advanced, Unresectable, or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000298994; ECOG-E1202
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Perifosine may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have locally advanced, unresectable, or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of perifosine, in terms of objective response, in patients with locally advanced, unresectable, or metastatic pancreatic cancer.
* Determine the response duration, progression-free survival, and overall survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral perifosine every 6 hours for a total of 6 doses and then once daily in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 35-84 patients will be accrued for this study within 21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas
* Locally advanced, unresectable, or metastatic disease
* Measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* AST no greater than 2 times upper limit of normal (ULN)
* Bilirubin no greater than 2 times ULN

Renal

* Creatinine no greater than 1.4 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for pancreatic cancer
* More than 6 months since prior chemotherapy for other diseases

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* At least 4 weeks since prior surgery and recovered

Other

* No other concurrent investigational agents for pancreatic cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert de W. Marsh, MD, Study Chair — University of Florida; Caio Max S. Rocha Lima, MD — H. Lee Moffitt Cancer Center and Research Institute
Locations (10):
- United States (10):
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Tufts - New England Medical Center, Boston, Massachusetts
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] Marsh Rde W, Rocha Lima CM, Levy DE, Mitchell EP, Rowland KM Jr, Benson AB 3rd. A phase II trial of perifosine in locally advanced, unresectable, or metastatic pancreatic adenocarcinoma. Am J Clin Oncol. 2007 Feb;30(1):26-31. doi: 10.1097/01.coc.0000251235.46149.43. PMID 17278891